CLINICAL TRIAL: NCT05902819
Title: An Investigation of the Effect of MMP-9 Inhibition With Minocycline on the Reconsolidation of Intrusive Trauma- or Cocaine-related Memories
Brief Title: Reconsolidation Blockade of Intrusive Trauma- and Cocaine-related Memories
Acronym: Memocycline
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022-01177
Record Dates: First submitted 2023-04-26; First posted 2023-06-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Post-traumatic Stress Disorder; Cocaine Use Disorder
Keywords: memory reconsolidation blockade; minocycline; MMP-9 inhibition; PTSD; cocaine use disorder; placebo-controlled
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel group, single center study
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- PTSD intervention group (Experimental): 30 individuals with PTSD will receive imagery with minocycline.
  Interventions: Behavioral: Imagery; Drug: Minocycline
- PTSD control group (Placebo Comparator): 30 individuals with PTSD will receive imagery with placebo.
  Interventions: Behavioral: Imagery; Drug: Placebo
- CUD intervention group (Experimental): 30 individuals with CUD will receive imagery with minocycline.
  Interventions: Behavioral: Imagery; Drug: Minocycline
- CUD control group (Placebo Comparator): 30 individuals with CUD will receive imagery with placebo.
  Interventions: Behavioral: Imagery; Drug: Placebo
- Healthy control group (No Intervention): 30 healthy individuals who will not receive any intervention.
- Clinical control group (No Intervention): 30 individuals with both PTSD and CUD who will not receive any intervention
- Healthy control group for memory narratives (No Intervention): 30 healthy individuals who will not receive any intervention, who undergo an online memory assessment only to improve comparability of text-based language features between healthy controls and participants with a PTSD or CUD diagnosis (HCN group)

INTERVENTIONS:
Behavioral: Imagery — Guided imagery of personal trauma- or cocaine-related memory approximately 120min after study medication was given.
  Arms: CUD control group; CUD intervention group; PTSD control group; PTSD intervention group
Drug: Minocycline — Single dose of minocycline (200mg) at each of two imagery sessions; Minocycline is given orally in form of a capsule.
  Arms: CUD intervention group; PTSD intervention group
Drug: Placebo — Single dose of mannitol (100%) at each of two imagery sessions; Placebo is given orally in form of a capsule.
  Arms: CUD control group; PTSD control group

SUMMARY:
An investigation of the effect of matrix-metalloproteinase-(MMP)-9 inhibition with minocycline on the reconsolidation of trauma- or cocaine-related memories

DETAILED DESCRIPTION:
Intrusive memories are involuntary recollections of past emotional events that can become pathological and persist over time, particularly in post-traumatic stress disorder (PTSD) and cocaine use disorders (CUD). Both PTSD and CUD are characterised by a hypersensitivity and -reactivity to cue-elicited memory reactivation and exhibit common neurological alterations, suggesting shared underlying mechanisms. As intrusive memories significantly contribute to maintaining the cycle of relapse in both disorders, it is important to find a way to attenuate them successfully. Research on memory reconsolidation has led to the development of different (pharmacological) approaches to disrupt the process, which have, however, yielded mixed and unspecific effects so far.

The present project aims to investigate the effect of MMP-9 inhibition with minocycline on the reconsolidation of intrusive memories in individuals with CUD or PTSD. Participants will be randomly assigned to a minocycline or placebo group. The study comprises a total of 5 visits during 3 weeks and one follow-up online survey (3 months after the intervention). Participants will receive the study medication before two imagery script-guided memory activation sessions. An ecological momentary assessment (EMA) approach will be employed to track intrusive memories, and glutamate concentration and neural activation will be measured with magnetic resonance spectroscopy (MRS) and functional magnetic resonance (fMRI), respectively, before and after the two imagery sessions.

ELIGIBILITY:
General Inclusion Criteria:

* Ability to read, understand and provide written informed consent
* Age between 18 and 60 years
* To be sufficiently fluent in German

Inclusion Criteria for the PTSD group:

- Current diagnosis of full PTSD according to the 5th version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), of subthreshold PTSD, as in meeting two to three of the DSM-5 criteria B-E, or of complex PTSD

Inclusion Criteria for the CUD group:

* Current diagnosis of mild, moderate, or severe CUD according to DSM-5
* Regular cocaine use in the last 12 months and at least one consumption event in the last 6 months

Inclusion Criteria for the Clinical Controls (PTSD+CUD group):

* Current diagnosis of full PTSD according to the 5th version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), of subthreshold PTSD, as in meeting two to three of the DSM-5 criteria B-E, or of complex PTSD
* Current diagnosis of mild, moderate, or severe CUD according to DSM-5
* Regular cocaine use in the last 12 months and at least one consumption event in the last 6 months

Exclusion Criteria for the HC, PTSD, CUD, and PTSD+CUD groups:

* Women who are pregnant or breast feeding or intending to become pregnant during the course of the study or within 3 months after
* Other clinically significant concomitant disease states, e.g., renal failure (i.e., estimated glomerular filtration rate (eGFR; CKD-EPI) lower than 60 ml/min/1.73 m2), hepatic dysfunction (i.e., alanine transaminase (ALT) higher than 90 U/I for women or 110 U/I for men, aspartate aminotransferase (AST) higher than 74 U/I, and/or gamma-glutamyl transferase (γGT) higher than 70 U/I for women or 120 U/I for men), cardiovascular disease, etc.
* Presence or history of severe neurological disorders, head injuries or systemic/rheumatic disease
* Diagnosis of schizophrenia, bipolar disorder, or autism spectrum disorder according to DSM-5
* Pacemaker, neurostimulator or any other head or heart implants as well as MRI-incompatible metal parts or possibility of metal fragments in the body (MR safety)
* Claustrophobia (MR safety)
* Dependence on a hearing aid (MR safety)
* Inability to follow the procedures of the study, e.g., due to language problems
* Participation in another study with investigational drugs within the 30 days preceding and during the present study
* More than three suicide attempts in the past, a suicide attempt within the last 12 months and/or acute suicidality

Exclusion Criteria for Healthy Controls:

* Any current psychiatric diagnosis according to DSM-5 except for mild or moderate substance use disorder (SUD) for nicotine, and mild SUD for alcohol and cannabis
* Diagnosis of CUD according to DSM-5 (lifetime)
* Diagnosis of PTSD according to DSM-5 (lifetime)

Exclusion Criteria for HCN:

* Any self-reported current psychiatric diagnosis except for mild or moderate SUD for nicotine (F17.2)
* Self-reported acute intoxication with alcohol or cannabis
* >25 intakes of cocaine, amphetamines, methamphetamine, MDMA, ketamine, psychedelics, benzodiazepines, other psychotropic substances such as novel psychoactive substances, non-prescribed opioids or methylphenidate
* Showing signs of acute mental health issues according to the GHQ-12 (Likert scale: cut-off 12 points)
* Self-reported suicidal ideations in the last 12 months

Exclusion Criteria for both the PTSD and CUD groups:

* Allergy to minocycline or to any other ingredient in the named drug
* Current intake of the following medications interacting with minocycline: acitretin, acetylcystein, aluminiumhydroxid, amitryptiline, any antibiotics, antidiabetic drug such as sulfonylurea, atazanavir, atomoxetine, anticoagulant drugs from the coumarin type, barbiturates, bupropion, carbamazepine, ciclosporin A, isotretinoin, methotrexate, phenytoin, and theophylline

Exclusion Criteria for only the PTSD group:

* Diagnosis of CUD according to DSM-5 (lifetime)
* Current diagnosis of severe SUD for nicotine, moderate SUD for alcohol and cannabis, and mild SUD for all other substances according to DSM-5

Exclusion Criteria for only the CUD group:

* Diagnosis of PTSD according to DSM-5 (lifetime)
* Current diagnosis of severe SUD for alcohol or cannabis, and mild SUD for all other substances (except for nicotine) according to DSM-5

Exclusion Criteria for Clinical Controls (PTSD+CUD group):

- Current diagnosis of severe SUD for alcohol or cannabis, and mild SUD for all other substances (except for nicotine) according to DSM-5

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Changes in intrusive memories frequency and features | Changes from baseline intrusive memories frequency and features after both 9 to 39 days (follow-up 1) and approx. 3.5 months (follow-up 2)
  Measured with the Intrusion Questionnaire, containing various items on intrusive memories frequency, arousal and distress as well as triggers, and responses.
Change over time in self-reported intrusive memories frequency, arousal and distress | EMA will be conducted for an average of 12 to 42 days (through study participation from baseline to 3 days after follow-up 1).
  Captured with a short version of the Intrusion Questionnaire implemented as smartphone-based ecological momentary assessment (EMA), containing items on arousal and distress from self-reported intrusive memories.
Changes in fMRI Blood-Oxygenation-Level Dependent (BOLD) contrasts | Changes from baseline fMRI BOLD contrasts after 9 to max. 39 days (follow-up 1).
  fMRI BOLD contrasts between conditions (neutral/stress/trauma for the PTSD group; neutral/reward/drug for the CUD group) and between groups.
Changes in MRS signal parameters | Change from baseline MRS-measured glutamate concentrations after 9 to max. 39 days (follow-up 1).
  Glutamate concentrations are measured using MRS in the amygdala in the PTSD group and in the nucleus accumbens in the CUD group.

SECONDARY OUTCOMES:
Change in heart rate variability (HRV) during fMRI memory reactivation | Change from baseline HRV after 9 to max. 39 days (follow-up 1).
  HRV will be measured during the fMRI cue-reactivity paradigm (listening to trauma- or cocaine-related narratives compared to trauma- and cocaine-unrelated narratives).
Change in respiratory rate during fMRI memory reactivation | Change from baseline respiratory rate after 9 to max. 39 days (follow-up 1).
  Respiratory rate will be measured during the fMRI cue-reactivity paradigm (listening to trauma- or cocaine-related narratives compared to trauma- and cocaine-unrelated narratives).
Change in subjective rating of distress before and after memory reactivation | Change from baseline subjective distress after 9 to max. 39 days (follow-up 1).
  Current subjective distress will be measured with a visual analogue scale before and after listening to trauma- and cocaine-related narratives compared to trauma- and cocaine-unrelated narratives.
Change in subjective rating of craving before and after memory reactivation | Change from baseline craving after 9 to max. 39 days (follow-up 1).
  Current subjective craving will be measured with the Cocaine Craving Questionnaire (containing ten questions on current craving scaled from 0 to 10) before and after listening to cocaine-related narratives compared to cocaine-unrelated narratives.
Change in neurofilament light chain (NfL) levels | Change from baseline NfL levels after 9 to max. 39 days (follow-up 1).
  NfL levels will be measured in serum samples.
Change in sphingolipid levels | Change from baseline sphingolipid levels after 9 to max. 39 days (follow-up 1).
  Sphingolipid levels will be measured in plasma samples.
Change in inflammatory biomarker levels | Change from baseline inflammatory levels after 9 to max. 39 days (follow-up 1).
  Inflammatory biomarker levels will be measured in serum samples.
Change in MMP-9 protein levels | Change from baseline MMP-9 protein levels after 9 to max. 39 days (follow-up 1).
  MMP-9 protein levels will be measured in plasma samples.
Change in MMP-9 gene expression | Change from baseline MMP-9 gene expression after 9 to max. 39 days (follow-up 1).
  MMP-9 gene expression will be measured in blood samples.
Heartrate variability | Will be measured during 9 to max. 39 days, from baseline until follow-up 1.
  Heartrate variability (measured with a wearable (Fitbit)) predicted by the number and quality of intrusive memories experienced. Overall variability per person, in relation to overall health measured at Screening and Baseline as well as pre- and post-intervention variability will be assessed.
Sleep duration | Will be measured during 9 to max. 39 days, from baseline until follow-up 1.
  Sleep duration (in minutes), trajectories over the course of the study periods, clusters of variations in duration and sleep quality (as averaged by the algorithm of Fitbit), according to medication/placebo, number of intrusions and overall health measured at Screening and Baseline.
Change in Obsessive Compulsive Cocaine Use Scale (OCCUS) | Change from baseline OCCUS score after both 9 to 39 days (follow-up 1) and approx. 3.5 months (follow-up 2).
  A 14-item self-report measure that assesses the current inability to control or resist cocaine-related thoughts and behaviors, frequency and impact of thoughts and impulses related to cocaine use, and the degree of interference caused by cocaine related thoughts and behaviors.
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline PCL-5 score after both 9 to 39 days (follow-up 1) and approx. 3.5 months (follow-up 2).
  A 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD in the last 2 weeks prior to the visit.
Beck Depression Inventory-II (BDI-II) | Change from baseline BDI-II score after both 9 to 39 days (follow-up 1) and approx. 3.5 months (follow-up 2).
  A 21-item self-report measure for assessing the severity of depression in the last 2 weeks prior to the visit.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline PSQI score after both 9 to 39 days (follow-up 1) and approx. 3.5 months (follow-up 2).
  A 19-item self-report measure which assesses sleep quality and disturbances in the last 2 weeks prior to the visit.
Global Assessment of Functioning (GAF) | Change from screening GAF score after both 10 to 50 days (follow-up 1) and approx. 4 months (follow-up 2).
  A numeric scale used by the investigators to rate the current social, occupational, and psychological functioning of a participants. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change from screening CAPS-5 score after approx. 4 months (follow-up 2).
  A 30-item structured interview that is used to assess the 20 DSM-5 PTSD symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since the previous CAPS administration, and overall PTSD severity, and specifications for the dissociative subtype.
Changes in the Interview for Psychotropic Drug Consumption (IPDC) | Change from screening IPDC after approx. 4 months (follow-up 2).
  A structured interview assessing self-reported patterns of use of common licit and illicit substances during the most representative month of the past year and, in the case of regular cocaine use, also specifically during the past month.
Voice-recorded language features of memories | Assessed at screening
  Voice features and text-based features of reported autobiographical memories recorded during the screening to predict symptoms, with a primary focus on the prediction of intrusion-related features.

CONTACTS AND LOCATIONS:
Overall Officials: Boris B. Quednow, Prof. Dr., Principal Investigator — Psychiatric University Hospital Zurich, University of Zurich; Birgit Kleim, Prof. Dr., Principal Investigator — Psychiatric University Hospital Zurich, University of Zurich
Locations (1):
- Psychiatric University Hospital Zurich, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No